CLINICAL TRIAL: NCT05602064
Title: Effectiveness of Pre-emptive Analgesics on Post-Operative Pain After Stainless Steel Crown Placement On Primary Molars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Farah Nemr, Instructor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 270221
Record Dates: First submitted 2022-10-18; First posted 2022-11-01 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Post-operative Pain
Keywords: Pre-emptive analgesia; ibuprofen; paracetamol; post-operative pain; stainless steel crown; Primary molars
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (Ibuprofen) (Experimental): Participants will receive ibuprofen 100 mg/5 ml (BRUFEN®, Kahira Pharmaceuticals & Chemical Industries Co.) The solution will be administered Once, 1 hour prior to the local anesthesia administration.
  The participant will receive a weight-dosed volume Effective dosages range from 10 mg/kg/day to a maximum of 40 mg/kg/day
  Interventions: Drug: Ibuprofen
- Group II (Paracetamol) (Experimental): Participants will receive paracetamol 250 mg/5 ml (CETAL®, EGYPTIAN INT. PHARMACEUTICAL INDUSTRIES CO.) The solution will be administered once, 1 hour prior to the local anesthesia administration.
  The participant will receive a weight-dosed volume Effective dosages are between 15-20mg/kg/day to a maximum of 60 mg/kg/day
  Interventions: Drug: Paracetamol
- Group III (Placebo) (Placebo Comparator): The placebo solution will be freshly prepared by an assistant in a manner to match the color and odor of the analgesics
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen is a non-steroidal anti-inflammatory drug which acts by reducing the production of cyclo-oxygenases (COX-1 and COX-2)- derived prostanoids in the blood
  Other Names: BRUFEN®, Kahira Pharmaceuticals & Chemical Industries Co.
  Arms: Group I (Ibuprofen)
Drug: Paracetamol — Paracetamol is an analgesic that acts peripherally; although its primary site of action is still debatable, it is thought to inhibit prostaglandins in the hypothalamus
  Other Names: CETAL®, EGYPTIAN INT. PHARMACEUTICAL INDUSTRIES CO.
  Arms: Group II (Paracetamol)
Other: Placebo — A placebo solution will be freshly prepared by an assistant in a manner to match the color and odor of the analgesics
  Arms: Group III (Placebo)

SUMMARY:
The aim of this study is to evaluate the effectiveness of pre-emptive analgesia using ibuprofen and paracetamol on reducing post-operative pain following the placement of stainless steel crowns on primary molars compared to placebo

DETAILED DESCRIPTION:
The study will be a parallel, placebo-controlled, triple-blinded, randomized clinical trial. A total of 66 healthy children aged 5-8 years requiring the placement of a stainless steel crown will be selected from Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Alexandria University, Egypt. The children will be randomly allocated into three groups according to the type of pre-emptive solution used. Group I will receive ibuprofen, group II will receive paracetamol, while group III (control) will receive a placebo solution. Children will self-report their level of pain using a Visual analogue scale (VAS) and/or a Facial pain scale (FPS) after local anesthesia administration, immediately after the cementation of the stainless steel crown, and 2, 6 and 24 hours post-operatively. Children's baseline anxiety and parental anxiety will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

Participant inclusion criteria:

* Age range 5 to 8 years old
* Children without any previous interventional dental experience
* Children free of any systemic disease or special health care needs (ASA 1)
* Children free of any allergies or hypersensitivity reactions to local anesthetics or analgesic drugs
* Positive or definitely positive behaviour during preoperative assessments according to the Frankl Rating Scale (score 3 or 4)
* Parents/caregivers and children who are willing to participate in the study

Tooth inclusion criteria:

* Maxillary first or second primary molar teeth with extensive and/or multisurface caries where other restorations are likely to fail but without pulp exposure
* Absence of clinical and radiographic signs or symptoms of irreversible pulpitis
* Absence of fistula or abscess near the selected tooth clinically and radiographically
* Absence of spontaneous pain
* Absence of pulp exposure
* Absence of pathological mobility by placing the points of a pair of tweezers in an occlusal fossa, and gently rocking the tooth bucco-lingually

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Post-operative pain evaluation | Day 0 (Immediately post-operatively)
  Pain will be measured via a visual analogue scale (VAS) based on a straight line of 100 mm where 0 mm indicates absence of pain and 100 mm indicates greatest pain felt, and a facial pain scale.Children will self-report their level of pain four times post-operatively
Post-operative pain evaluation | Day 0 (2 hours post-operatively)
  Pain will be measured via a visual analogue scale (VAS) based on a straight line of 100 mm where 0 mm indicates absence of pain and 100 mm indicates greatest pain felt, and a facial pain scale.Children will self-report their level of pain four times post-operatively
Post-operative pain evaluation | Day 0 (6 hours post-operatively)
  Pain will be measured via a visual analogue scale (VAS) based on a straight line of 100 mm where 0 mm indicates absence of pain and 100 mm indicates greatest pain felt, and a facial pain scale.Children will self-report their level of pain four times post-operatively
Post-operative pain evaluation | Day1 (24 hours post-operatively)
  Pain will be measured via a visual analogue scale (VAS) based on a straight line of 100 mm where 0 mm indicates absence of pain and 100 mm indicates greatest pain felt, and a facial pain scale.Children will self-report their level of pain four times post-operatively

SECONDARY OUTCOMES:
Trans-operative pain evaluation | Day 0 (During Procedure)
  To assess the effectiveness of pre-emptive analgesics in reducing pain during local anesthesia administration, after local anesthesia administration, the child will be shown the Visual analogue scale (VAS) based on a straight line of 100 mm where 0 mm indicates absence of pain and 100 mm indicates greatest pain felt, and a Facial Pain Scale (FPS). He/she will be asked to choose the score or face which best describes the level he/she felt during administration of the anesthetic solution.
Evaluation of the child's dental anxiety | Day0 (In the waiting room before the intervention)
  To assess the child's anxiety, the Arabic version of the faces version of Modified Child Dental Anxiety Scale (MCDASf) will be used.The MCDAS consists of eight questions to assess dental anxiety about specific dental procedures. A five-point Likert scale is used to determine dental anxiety with scores ranging from 'relaxed/not worried' to 'very worried'. The faces version of Modified Child Dental Anxiety Scale (MCDASf) has a faces analogue scale anchored above the original numeric form.
Evaluation of parental anxiety | Day 0 (In the waiting room before the intervention)
  Parental anxiety will be evaluated using the Arabic version of the Modified Dental Anxiety Scale (MDAS) which consists of 5 questions with a score of 0 to 4, where 0 indicates absence of anxiety and 4 indicates being extremely anxious.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Dentistry department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT05602064/Prot_SAP_000.pdf